CLINICAL TRIAL: NCT02420431
Title: Improving the Effectiveness of Psychological Interventions for Depression and Anxiety in the Cardiac Rehabilitation Pathway: A Single-blind Randomised Controlled Trial
Brief Title: Treating Depression and Anxiety in the Cardiac Rehabilitation Pathway
Acronym: PATHWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Manchester Mental Health & Social Care Trust (Other Government); University of Liverpool (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical and Experimental Psychopathology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156862 (RP-PG-1211-20011)
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety; Cardiac Rehabilitation
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cardiac Rehabilitation; Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metacognitive therapy plus CR (Experimental): Group psychological treatment focused on reducing worry and rumination and modifying beliefs about thinking in addition to treatment as usual (standard cardiac rehabilitation)
  Interventions: Behavioral: Metacognitive Therapy
- CR alone (control) (Active Comparator): Usual group-based cardiac rehabilitation (treatment as usual) involving stress management, exercise, education
  Interventions: Behavioral: Cardiac Rehabilitation (treatment as usual)

INTERVENTIONS:
Behavioral: Metacognitive Therapy — Metacognitive therapy (MCT) helps clients to identify episodes of worry and rumination in response to negative thoughts and bring these responses under control. This process is facilitated by exercises that enhance the flexibility of attention control, challenge unhelpful beliefs about thinking and enable new relationships with thoughts
  Arms: metacognitive therapy plus CR
Behavioral: Cardiac Rehabilitation (treatment as usual) — Stress management, relaxation training, exercise and dietary advice.
  Arms: CR alone (control)

SUMMARY:
Cardiac rehabilitation (CR) services aim to improve heart disease patients' health and quality of life, and reduce the risk of further cardiac events. Depression and anxiety (distress) are common among CR patients: 37% of patents have significant anxiety and/or depressive symptoms. Distressed patients are at greater risk of death, further cardiac events and poorer quality of life than those without distress and they use more healthcare. Available drug and psychological treatments have only small effects on distress and quality of life, and no effects on physical health. Therefore, it is essential that more effective treatments for depression and anxiety are integrated into CR services. Extensive evidence shows that a particular style of thinking dominated by rumination (dwelling on the past) and worry maintains emotional distress. A psychological intervention (metacognitive therapy) that reduces this style of thinking alleviates depression and anxiety in mental health settings. The investigators aim to conduct a pilot trial of the group intervention and in work stream 2 the investigators will undertake a full-scale trial to evaluate whether adding the group intervention to standard CR is more effective at alleviating anxiety and depression than standard CR alone.

ELIGIBILITY:
Inclusion Criteria:

* Heart disease patients referred to CR with: Acute coronary syndrome
* Following revascularisation; stable heart failure
* Stable angina, implanted cardioverter defibrillators
* Heart valve repair/replacement
* Heart transplantation and ventricular assist devices
* Adult congenital heart disease
* Must have a score of 8 or more on either the depression or anxiety subscale of the HADS
* Competent level of English language skills

Exclusion Criteria:

* Cognitive impairment which precludes informed consent/ability to participate
* Acute suicidality
* Active psychotic disorders
* Current drug/alcohol abuse
* Concurrent psychological intervention for emotional distress
* Antidepressant or anxiolytic medication initiated in previous 8 weeks
* Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2015-07; Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline pre treatment, four-month post baseline

SECONDARY OUTCOMES:
Impact of Events Scale -revised | Baseline, four-month post baseline, 12 months follow-up
Metacognitions Questionnaire 30 | Baseline, four-month post baseline, 12 month follow-up
Cognitive Attentional Syndrome scale (CAS-1) | Baseline, four-month post baseline, 12 months follow-up
Health Related Quality of Life (EQ-5D) | Baseline, four-month post baseline, 12 months follow-up
Economic Patient Questionnaire | Baseline, 4 month follow-up, 12 months follow-up
Hospital Anxiety and Depression Scale | 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, Ph.D, Principal Investigator — University of Manchester
Locations (5):
- United Kingdom (5):
  - Macclesfield District General Hospital, Macclesfield, Cheshire
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, Lancashire
  - University Hospital of South Manchester NHS Foundation Trust, Manchester, Lancashire
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Stepping Hill Hospital, Manchester

REFERENCES:
- [Result] Wells A, Reeves D, Capobianco L, Heal C, Davies L, Heagerty A, Doherty P, Fisher P. Improving the Effectiveness of Psychological Interventions for Depression and Anxiety in Cardiac Rehabilitation: PATHWAY-A Single-Blind, Parallel, Randomized, Controlled Trial of Group Metacognitive Therapy. Circulation. 2021 Jul 6;144(1):23-33. doi: 10.1161/CIRCULATIONAHA.120.052428. Epub 2021 Jun 21. PMID 34148379
- [Derived] Wells A, Reeves D, Heal C, Davies LM, Shields GE, Heagerty A, Fisher P, Doherty P, Capobianco L. Evaluating Metacognitive Therapy to Improve Treatment of Anxiety and Depression in Cardiovascular Disease: The NIHR Funded PATHWAY Research Programme. Front Psychiatry. 2022 Jun 3;13:886407. doi: 10.3389/fpsyt.2022.886407. eCollection 2022. PMID 35722590
- [Derived] McPhillips R, Salmon P, Wells A, Fisher P. Cardiac Rehabilitation Patients' Accounts of Their Emotional Distress and Psychological Needs: A Qualitative Study. J Am Heart Assoc. 2019 Jun 4;8(11):e011117. doi: 10.1161/JAHA.118.011117. Epub 2019 Jun 1. PMID 31433708